CLINICAL TRIAL: NCT00711802
Title: An Evaluation of the Safety, Efficacy and Pharmacokinetics of Daptomycin in Pediatric Subjects Aged One to Seventeen Years With Complicated Skin and Skin Structure Infections Caused by Gram-Positive Pathogens
Brief Title: Safety and Efficacy Study of Daptomycin in Pediatric Participants (1 to 17 Years-old) With Skin and Skin Structure Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3009-017; DAP-PEDS-07-03 (Other: Cubist Study Number)
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Skin Diseases, Infectious
Keywords: Complicated; Skin; Structure
MeSH Terms: conditions — Skin Diseases, Infectious | interventions — Daptomycin; Standard of Care; Nafcillin; Oxacillin; Cloxacillin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daptomycin (Experimental): Administered intravenously (IV) every 24 hours for up to 14 days at the following age-dependent dosages.
  Participants ages 7 to 17 years: daptomycin was dissolved in a volume of 50 milliliters (mL) 0.9% sodium chloride for injection over 30 minutes (min) with an infusion rate of 1.67 mL/min.
  Participants 1 to 6 years-old: daptomycin was dissolved in a volume of 25 mL 0.9% sodium chloride for injection over 60 min with an infusion rate was 0.42 mL/min.
  Age Group 1 (for ages 12 to 17 years): 5 milligrams/kilogram (mg/kg)
  Age Group 2 (for ages 7 to 11 years): 7 mg/kg
  Age Group 3 (for ages 2 to 6 years): 9 mg/kg
  Age Group 4 (for ages 1 to <2 years): 10 mg/kg
  Interventions: Drug: Daptomycin
- Standard of Care (SOC) (Active Comparator): The comparator agent for this study was the SOC treatment and dosage deemed appropriate by the Investigator. The recommended SOC agents were IV vancomycin, IV clindamycin, and IV semisynthetic penicillins every 24 hours for up to 14 days.
  Interventions: Drug: Standard of Care (SOC)

INTERVENTIONS:
Drug: Daptomycin
  Other Names: Cubicin
  Arms: Daptomycin
Drug: Standard of Care (SOC)
  Other Names: nafcillin, oxacillin, cloxacillin
  Arms: Standard of Care (SOC)

SUMMARY:
This is a multi-center, evaluator-blinded, randomized, comparative study designed to assess the safety, efficacy, and pharmacokinetics (PK) of daptomycin in pediatric subjects ages 1 to 17 years, inclusive, with complicated skin and skin structure infections (cSSSI) caused by Gram-positive pathogens.

DETAILED DESCRIPTION:
This is a multi-center, evaluator-blinded, randomized, comparative study designed to assess the safety, efficacy, and PK of daptomycin in pediatric participants ages 1 to 17 years, inclusive, with cSSSI caused by Gram-positive pathogens. Participants will be enrolled into age groups and given age-dependent doses over a period of up to 14 days. Participants will be stratified by age group to receive either daptomycin or SOC (recommended as vancomycin, clindamycin or semisynthetic penicillin) in a ratio of 2:1, respectively. Participants may continue on oral therapy following completion of IV study drug administration and provided that the participant meets all criteria for conversion to oral therapy, including clear clinical improvement and availability of an oral agent to which the pathogen is susceptible. The choice of oral therapy will be left to the discretion of the Investigator. February 11, 2015 released from post marketing requirement to include subjects aged 3 months - < 1 year. Ref ID: 3701325

ELIGIBILITY:
Inclusion Criteria:

* Written parental (or appropriate legal representative) informed consent prior to any study-related procedure not part of normal medical care
* Written participant assent (as appropriate)
* Male or female between the ages of 1 and 17 years old, inclusive
* If female of childbearing potential (defined as post-menarche), not lactating or pregnant, documented negative pregnancy test result within 48 hours prior to study medication administration and willing to practice reliable birth control measures (at the discretion of the Principal Investigator) during study treatment and for at least 28 days after study completion
* Able to comply with the protocol for the duration of the study
* Skin and skin structure infections of a complicated nature known or suspected to be caused by Gram-positive pathogen(s) that require IV antibiotic treatment. Complicated infections are defined as infections either involving deep soft tissue or requiring significant surgical intervention (such as, infected ulcers, burns, and major abscesses) or infections in which the participant has a significant underlying disease state that complicates the response to treatment. The Investigator may contact the Medical Monitor to discuss infections not meeting this definition but which otherwise appear appropriate for inclusion
* At least three of the following clinical signs and symptoms associated with the cSSSI: pain; tenderness to palpation; temperature >37.5 degrees Celsius (C) (99.5 degrees Fahrenheit [F]) oral or >38 degrees C (100.4 degrees F) rectal; white blood count (WBC) >12,000/cubic millimeter (mm^3) or ≥10% bands; swelling and/or induration; erythema (>1 centimeter [cm] beyond edge of wound or abscess); or pus formation

Exclusion Criteria:

* Investigational drug use (including daptomycin) or participation in any experimental procedure in the 30 days preceding study entry
* Known allergy/hypersensitivity to daptomycin
* Known infection caused solely by Gram-negative pathogen(s), fungus(i), or virus(es)
* Previous systemic antimicrobial therapy exceeding 24 hours in duration administered anytime during the 48 hours prior to the first dose of study drug (exception: a participant is eligible if on previous antibiotics without any clinical improvement and/or a wound culture is available and the pathogen is not sensitive to prior therapy)
* Known or suspected pneumonia, osteomyelitis, meningitis, or endocarditis
* Known bacteremia (exception: any participant enrolled in the study that is subsequently found to have a blood culture positive for bacteremia may be continued)
* Participant with current or known clinically significant abnormal laboratory test results (including electrocardiograms [ECGs]) that would expose the participant to unacceptable risk as determined by Investigator
* History of clinically significant cardiovascular, renal, hepatic, pulmonary (well-controlled asthma is acceptable), gastrointestinal, endocrine, hematological, autoimmune disease, or primary immune deficiency (unless the Investigator considers that the subject would not be at risk by participating in the study [Note: human immunodeficiency virus-infected participants must not be enrolled])
* History of or current clinically significant (at the discretion of the Investigator) muscular disease, nervous system, or seizure disorder
* Unexplained muscular weakness, history of peripheral neuropathy, Guillain-Barre syndrome or spinal cord injury
* Known or suspected renal insufficiency (that is, estimated creatinine clearance rate [CLcr]<80 mL/min/1.73 squared meter [m^2]
* History of or current rhabdomyolysis
* History of (within 1 year prior to first dose of study drug) or current myositis
* Current septic shock
* Known or suspected creatine phosphokinase (CPK) elevation

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 396 (Actual)
Dates: Start 2008-07-23 (Actual); Primary Completion 2013-10-11 (Actual); Study Completion 2013-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Hershberger, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (30):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of South Florida College of Medicine, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Montifiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - LeBonheur Children's Medical Center, Memphis, Tennessee
  - Vanderbilt University Medical Center and Children's Hospital, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas Health Science Center, Houston, Texas
- India (7):
  - Medisys Hospital, Bangalore
  - MS Ramaiah, Bangalore
  - MV Hospital and Research Center, Lucknow
  - BYL Nair Hospital, Mumbai
  - Lokmanya Tilak Municipal Medical College, Mumbai
  - KEM Hospital, Pune
  - Ruby Hall Clinic, Pune
- Hospital Del Nino, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Bradley J, Glasser C, Patino H, Arnold SR, Arrieta A, Congeni B, Daum RS, Kojaoghlanian T, Yoon M, Anastasiou D, Wolf DJ, Bokesch P. Daptomycin for Complicated Skin Infections: A Randomized Trial. Pediatrics. 2017 Mar;139(3):e20162477. doi: 10.1542/peds.2016-2477. Epub 2017 Feb 15. PMID 28202770

RESULTS

PARTICIPANT FLOW:
Groups:
- Age Group 1: Daptomycin: Daptomycin: 5 milligrams/kilogram (mg/kg) administered intravenously (IV) every 24 hours for up to 14 days
  Age Group 1: Participants ages 12 to 17 years
- Age Group 1: Standard of Care (SOC): SOC: The comparator agent for this study was the SOC treatment and dosage deemed appropriate by the Investigator. The recommended SOC agents were IV vancomycin, IV clindamycin, and IV semisynthetic penicillins every 24 hours for up to 14 days.
  Age Group 1: Participants ages 12 to 17 years
- Age Group 2: Daptomycin: Daptomycin: 7 mg/kg administered IV every 24 hours for up to 14 days
  Age Group 2: Participants ages 7 to 11 years
- Age Group 2: SOC: SOC: The comparator agent for this study was the SOC treatment and dosage deemed appropriate by the Investigator. The recommended SOC agents were IV vancomycin, IV clindamycin, and IV semisynthetic penicillins every 24 hours for up to 14 days.
  Age Group 2: Participants ages 7 to 11 years
- Age Group 3: Daptomycin: Daptomycin: 9 mg/kg administered IV every 24 hours for up to 14 days
  Age Group 3: Participants ages 2 to 6 years
- Age Group 3: SOC: SOC: The comparator agent for this study was the SOC treatment and dosage deemed appropriate by the Investigator. The recommended SOC agents were IV vancomycin, IV clindamycin, and IV semisynthetic penicillins every 24 hours for up to 14 days.
  Age Group 3: Participants ages 2 to 6 years
- Age Group 4: Daptomycin: Daptomycin: 10 mg/kg administered IV every 24 hours for up to 14 days
  Age Group 4: Participants ages 1 to <2 years
- Age Group 4: SOC: SOC: The comparator agent for this study was the SOC treatment and dosage deemed appropriate by the Investigator. The recommended SOC agents were IV vancomycin, IV clindamycin, and IV semisynthetic penicillins every 24 hours for up to 14 days.
  Age Group 4: Participants ages 1 to <2 years
Period: Overall Study
Arm/Group | Age Group 1: Daptomycin | Age Group 1: Standard of Care (SOC) | Age Group 2: Daptomycin | Age Group 2: SOC | Age Group 3: Daptomycin | Age Group 3: SOC | Age Group 4: Daptomycin | Age Group 4: SOC
Started | 75 | 38 | 75 | 38 | 83 | 42 | 30 | 15
Received at Least 1 Dose of Study Drug | 73 | 37 | 73 | 38 | 81 | 42 | 30 | 15
Completed | 73 | 32 | 69 | 35 | 69 | 34 | 25 | 13
Not Completed | 2 | 6 | 6 | 3 | 14 | 8 | 5 | 2
Not completed — Not treated (no further detail) | 2 | 1 | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Microbiological failure | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1 | 10 | 6 | 4 | 2
Not completed — Reason not reported | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Age Group 1: Daptomycin: Daptomycin: 5 mg/kg administered IV every 24 hours for up to 14 days
  Age Group 1: Participants ages 12 to 17 years
- Total: Total of all reporting groups
Arm/Group | Age Group 1: Daptomycin | Age Group 1: Standard of Care (SOC) | Age Group 2: Daptomycin | Age Group 2: SOC | Age Group 3: Daptomycin | Age Group 3: SOC | Age Group 4: Daptomycin | Age Group 4: SOC | Total
Number analyzed (Participants) | 73 | 37 | 73 | 38 | 81 | 42 | 30 | 15 | 389
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.02 (1.584) | 14.84 (1.735) | 9.05 (1.443) | 8.98 (1.305) | 3.92 (1.556) | 3.86 (1.555) | 1.46 (0.299) | 1.43 (0.299) | 8.21 (5.134)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 15 | 28 | 15 | 48 | 20 | 21 | 12 | 188
  Male | 44 | 22 | 45 | 23 | 33 | 22 | 9 | 3 | 201
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 33 | 16 | 49 | 25 | 1 | 0 | 0 | 1 | 125
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 6 | 8 | 5 | 33 | 10 | 12 | 4 | 90
  White | 28 | 14 | 15 | 7 | 43 | 31 | 18 | 9 | 165
  More than one race | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any treatment-emergent adverse event (AE) that occurred from the time of first dose of the study drug through the last study evaluation or pre-existing adverse AEs that were aggravated in severity or frequency during the dosing period. The percentage of participants with at least 1 TEAE, with at least one drug-related AE (drug-related included "possibly related" or "related" as deemed by the Investigator; it also included events if causality was missing), and who discontinued from treatment due to a TEAE is presented. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 14 days after last dose of study drug
Population: Participants who received at least 1 dose of study drug with evaluable post-baseline TEAE data.
Measure: Number; unit: percentage of participants
Arm/Group | Age Group 1: Daptomycin | Age Group 1: Standard of Care (SOC) | Age Group 2: Daptomycin | Age Group 2: SOC | Age Group 3: Daptomycin | Age Group 3: SOC | Age Group 4: Daptomycin | Age Group 4: SOC
Number analyzed (Participants) | 72 | 38 | 73 | 38 | 81 | 42 | 30 | 15
percentage of participants
  At least 1 TEAE | 36.1 | 36.8 | 23.3 | 18.4 | 50.6 | 38.1 | 46.7 | 73.3
  At least 1 drug-related TEAE | 13.9 | 10.5 | 5.5 | 10.5 | 22.2 | 21.4 | 10.0 | 33.3
  Discontinued treatment due to a TEAE | 2.8 | 0 | 1.4 | 0 | 3.7 | 14.3 | 3.3 | 6.7

2. Secondary Outcome: Percentage of Participants With an Overall Therapeutic Response at Test of Cure Visit
Description: The assessment of therapeutic response was determined by comparing a participant's signs and symptoms at the test of cure visit (up to 14 days after last dose) to those recorded at baseline. Participants were classified as "Success" or "Failure" by combining their clinical and microbiological efficacy responses. Resolution of clinically significant signs and symptoms associated with the skin infection present at study baseline was considered "Success" by the Investigator. These participants were deemed both clinically cured and microbiologically eradicated. For participants whose clinical course could not be clearly defined as improved, a clinical outcome of "Failure" was rendered. In addition, if it was determined that the primary site of infection required additional antibiotic treatment, the assessment of clinical response was "Failure." If the Investigator was unable to determine a response because the participant was lost to follow-up, the assessment was "Unable to evaluate."
Time Frame: Baseline through 14 days after last dose of study drug
Population: Participants who received at least 1 dose of study drug with evaluable test-of-cure visit data.
Measure: Number; unit: percentage of participants
Arm/Group | Age Group 1: Daptomycin | Age Group 1: Standard of Care (SOC) | Age Group 2: Daptomycin | Age Group 2: SOC | Age Group 3: Daptomycin | Age Group 3: SOC | Age Group 4: Daptomycin | Age Group 4: SOC
Number analyzed (Participants) | 73 | 37 | 73 | 38 | 81 | 42 | 30 | 15
percentage of participants
  Clinical success | 95.9 | 91.9 | 90.4 | 92.1 | 82.7 | 76.2 | 80.0 | 86.7
  Clinical failure | 0 | 2.7 | 2.7 | 0 | 1.2 | 0 | 0 | 0
  Unable to evaluate | 4.1 | 5.4 | 6.9 | 7.9 | 16.1 | 23.8 | 20.0 | 13.3

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration-Time Curve for Daptomycin From 0 to the Last Sampling Time Point (AUC[0-t])
Description: Participants who volunteered for PK sampling had a blood sample collected for analysis at the following time points:
  Age Group 1; Day 3: Predose, 0.25 hour (hr), 1 hr, 4 hr, and12 hr postdose. Age Group 2; Day 3: Predose, 0.25 hr, 1 hr, 6 hr, and 10 hr postdose. Age Group 3; Day 1, 2, or 3: Predose, 0.25 hr, 1 hr, 6 hr, and 8 hr postdose. Age Group 4; Day 1, 2, or 3: 0, 1, 2, 4, and 6 hr relative to end of infusion.
Time Frame: Predose and 5 timepoints according to age group (up to 12 hours postdose)
Population: Participants who received at least 1 dose of study drug with evaluable daptomycin AUC(0-t) data.
Measure: Mean (Standard Deviation); unit: microgram*hour per milliliter (μg*hr/mL)
Arm/Group | Age Group 1: Daptomycin | Age Group 2: Daptomycin | Age Group 3: Daptomycin | Age Group 4: Daptomycin
Number analyzed (Participants) | 6 | 2 | 7 | 30
microgram*hour per milliliter (μg*hr/mL) | 318 (62.2) | NA (NA) — Due to limited pharmacokinetic (PK) samples, these measures could not be calculated. | 318 (68.6) | 466 (NA) — Due to limited PK samples, PK parameters were computed using the mean concentration-time profile during a sampling interval. As a result, no variability could be calculated.

ADVERSE EVENTS:
Time Frame: Baseline through 14 days after last dose of study drug
Description: Participants who received at least 1 dose of study drug with evaluable post-baseline TEAE data are included. Participants who experience more than one event are counted only once per System Organ Class and Preferred Term.
Arm/Group | Age Group 1: Daptomycin | Age Group 1: Standard of Care (SOC) | Age Group 2: Daptomycin | Age Group 2: SOC | Age Group 3: Daptomycin | Age Group 3: SOC | Age Group 4: Daptomycin | Age Group 4: SOC
Serious Adverse Events (participants affected / at risk) | 3/72 | 1/38 | 1/73 | 1/38 | 2/81 | 1/42 | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 15/72 | 9/38 | 7/73 | 2/38 | 27/81 | 10/42 | 11/30 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group 1: Daptomycin (N=72) | Age Group 1: Standard of Care (SOC) (N=38) | Age Group 2: Daptomycin (N=73) | Age Group 2: SOC (N=38) | Age Group 3: Daptomycin (N=81) | Age Group 3: SOC (N=42) | Age Group 4: Daptomycin (N=30) | Age Group 4: SOC (N=15)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic shock syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group 1: Daptomycin (N=72) | Age Group 1: Standard of Care (SOC) (N=38) | Age Group 2: Daptomycin (N=73) | Age Group 2: SOC (N=38) | Age Group 3: Daptomycin (N=81) | Age Group 3: SOC (N=42) | Age Group 4: Daptomycin (N=30) | Age Group 4: SOC (N=15)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 12 (13) | 4 (4) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 2 (3) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida nappy rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 8 (8) | 2 (2) | 1 (1) | 2 (2)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte percentage increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cells urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days